CLINICAL TRIAL: NCT02418052
Title: Effect of Neck Flexion on Post-operative Esophagogastric Anastomotic Leakage After Minimally Invasive Esophagectomy: a Single-center Randomized Controlled Trial
Brief Title: Effect of Neck Flexion on Esophagogastric Anastomotic Leakage After MIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Kun Li, MD, Kun Li, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kli2
Record Dates: First submitted 2015-04-12; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Esophageal Neoplasms; Esophagectomy; Anastomotic Leak
Keywords: esophageal cancer; minimally invasive esophagectomy; anastomotic leak; neck flexion
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neck flexion group (Experimental): Patients who fixed in neck flexion position after MIE
  Interventions: Procedure: neck flexion
- control group (No Intervention): Patients without posture intervention after MIE

INTERVENTIONS:
Procedure: neck flexion — After the cervical esophagogastric anastomoses is completed and the skin incision is closed, the patient's occiput will be lifted, and then the neck will be maintained in flexing position by an assistant. The underside of the chin will be fixed to the anterior chest wall with two stout nylon sutures by the surgeon. The neck will be fixed in the neutral flexing position for 7 to 10 days after surgery.
  Arms: neck flexion group

SUMMARY:
Esophageal cancer (EC) is the eighth most common cancer and the sixth leading cause of cancer deaths worldwide. Minimally invasive esophagectomy (MIE) is regarded as a safe and effective management for resectable EC. Gastric tube is considered to be an ideal substitute for the resected esophagus, and used for cervical esophagogastric anastomoses for digestive tract reconstruction in MIE. However, the tension at the anastomosed area can not be ignored and may cause cervical anastomotic leakage (CAL) in some cases. Continuous neck flexion is a standard post-operative posture after tracheal resection and reconstruction, and aimed to relieve the anastomotic tension. In this study, the investigators attempt to adopt the maneuver in MIE, and observe its effect on relieving the anastomotic tension and decreasing the incidence of CAL.

DETAILED DESCRIPTION:
After the cervical esophagogastric anastomoses is completed and the skin incision is closed, the patient's occiput will be lifted, and then the neck will be maintained in flexing position by an assistant. The underside of the chin will be fixed to the anterior chest wall with two stout nylon sutures by the surgeon. The neck will be fixed in the neutral flexing position for 7 to 10 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma of the intrathoracic esophagus.
* Surgical resectable (T1-4a, N0-3, M0).
* Age≥18 and ≤75 years.
* European Clinical Oncology Group (ECOG) performance status 0,1 or 2.
* Written informed consent obtain.

Exclusion Criteria:

* Carcinoma of the cervical esophagus.
* Carcinoma of the gastro-esophageal junction (GEJ).
* Prior thoracic surgery or trauma on the right hemithorax, or previous diseases which may lead to right pleural adhesion (these patients will undergo open surgery instead of minimally invasive esophagectomy). -Dysfunction of cardiorespiratory system or other surgical contraindications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative cervical esophagogastric anastomotic leakage | From the day of operation to hospital discharge (an expected average of 2 weeks)
  The post-operative cervical esophagogastric anastomotic leakage is defined as a radiological defect at the anastomotic site, or leakage of swallowed fluid (saliva, gastric juice or food residue) out of the drain site or cervical wound.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Li, MD, Study Chair — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China